CLINICAL TRIAL: NCT05957250
Title: [68Ga]Ga-FAPI-46 Positron Emission Tomography in Pancreaticobiliary Cancers: a Pharmacokinetics, Repeatability and Diagnostic Accuracy Study
Brief Title: [68Ga]Ga-FAPI-46 Positron Emission Tomography (PET) Scan to Improve the Imaging of Pancreatic and Bile Duct Cancer
Acronym: PANSCAN-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Dutch Cancer Society (Other); Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Dr. R.J. (Rutger-Jan) Swijnenburg, Principal Investigator, Oncological Surgeon, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL81511.018.22; 2022-001867-29 (EudraCT Number); 2022.0640 (Other: MERC approval number)
Record Dates: First submitted 2023-01-25; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Pancreatic Cancer; Cholangiocarcinoma
Keywords: Positron Emission Tomography; PET/CT; FAPI; Fibroblast activation protein; Radiopharmaceuticals
MeSH Terms: conditions — Pancreatic Neoplasms; Cholangiocarcinoma

STUDY DESIGN:
Intervention Model Description: Monocenter, non-randomized, non-blinded, prospective observational study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [68Ga]Ga-FAPI-46 PET/CT (Experimental): Depending on study fase: injection(s) with [68Ga]Ga-FAPI-46 for one or two [68Ga]Ga-FAPI-46 PET/CT scan(s)
  Interventions: Diagnostic Test: [68Ga]Ga-FAPI-46 PET/CT

INTERVENTIONS:
Diagnostic Test: [68Ga]Ga-FAPI-46 PET/CT — one or two [68Ga]Ga-FAPI-46 PET/CT scan(s)

SUMMARY:
The goal of this clinical trial is to evaluate the clinical use of [68Ga]Ga-FAPI-46 PET (positron emission tomography)/CT (computed tomography) imaging in patients with pancreatic or bile duct cancer. The study consists of three parts and patients can only participate in one part of the study.

The main questions the study aims to answer are:

* In part A: What is the best timing and scanprotocol of a [68Ga]Ga-FAPI-46 PET/CT scan?
* In part B: Are the results of the simplified scan protocol repeatable?
* In part C: What is the accuracy of [68Ga]Ga-FAPI-46 PET/CT to detect pancreatic cancer and is it able to detect the effect of chemotherapy on pancreatic cancer lesions?

Participants in this study will be asked to undergo the following:

* In part A: participants will undergo 1 [68Ga]Ga-FAPI-46 PET/CT scan and will have 2 venous canullas and 1 arterial cannula placed.
* In part B: participants will undergo 2 [68Ga]Ga-FAPI-46 PET/CT scans and will have a venous cannula placed for each scan.
* In part C: participants will undergo 2 [68Ga]Ga-FAPI-46 PET/CT scans and will have a venous cannula placed for each scan.

DETAILED DESCRIPTION:
Pancreaticobiliary cancer patients have a dismal prognosis. Therefore, patient stratification for the proper primary treatment is crucial to prevent unnecessary surgery and opens up the opportunity for novel (multimodal) treatment. Unfortunately, conventional imaging modalities are not sensitive enough to detect small tumor lesions or differentiate between benign and malignant tissue after neoadjuvant therapy. Tumor-specific imaging, using PET/CT imaging, can identify tumor tissue more accurately and therefore can improve lesion detection and patient stratification. Fibroblast activation protein (FAP) shows promise as a target to identify pancreaticobiliary cancers, lymph node metastases, and residual disease after neoadjuvant therapy. The FAP targeted inhibitor (FAPI) is developed to target FAP and has been labelled to the Gallium-68 (68Ga) radioisotope, resulting in the [68Ga]Ga-FAPI-46 tracer.

This study will be a three part monocenter study focusing on the clinical evaluation of [68Ga]Ga-FAPI-46.

* In part A, the pharmacokinetics of this tracer will be studied and the simplified method(s) to quantify tracer uptake will be validated.
* In part B, a test-retest study will be performed to assess the repeatability of these simplified quantitative methods.
* In part C, the sensitivity and feasibility of therapy response monitoring will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* Before patient registration, written informed consent must be given according to ICH/GCP, and national/local regulations.
* Additional Part A: patients with pancreaticobiliary cancer (pancreatic, intra- or extrahepatic cholangiocarcinoma) and a tumor size of >20mm on CT.
* Additional Part B: patients with primary pancreatic (or pancreaticobiliary) cancer (depending on the results of part A) and a tumor size of >20mm on CT. No treatment may be given in between the two scans.
* Additional Part C: patients with pathologically proven pancreatic ductal adenocarcinoma, eligible for neoadjuvant therapy before surgical resection.

Exclusion Criteria:

* Women who are pregnant and/or lactating.
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent. Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
* Impaired renal function (creatinine clearance <60 mL/min according to the Cockcroft-Gault equation.
* Leucocytes (WBC) ≤3.0 x 10^9/l
* Platelets ≤ 100 x 10^9 /l
* Hemoglobin ≤ 6 mmol/l
* Known hypersensitivity to drugs comparative to [68Ga]Ga-FAPI-46, or any of the excipients of [68Ga]Ga-FAPI-46.
* Inability to undergo PET/CT scanning (e.g. claustrophobia, weight limits or inability to tolerate lying for the duration of a PET/CT scan (~90 min)).

Additional Part A:

• Contra-indication for arterial cannula (e.g. inadequate circulation of extremity, positive Allen test, severe atherosclerosis, coagulant disorder (INR >1.4 or APTT >50)).

Additional Part C:

* Not eligible for surgery after neoadjuvant chemotherapy.
* If based on the first FAPI-46 PET/CT, there is a suspicion of metastatic disease the images will be discussed in the multidisciplinary meeting and one additional imaging modality (and a biopsy, if this would lead to a change of treatment strategy) can be used to confirm the suspicion. If metastatic disease is confirmed the patient will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Semi quantitative measurements of [68Ga]Ga-FAPI-46 tracer | 3 months
  [68Ga]Ga-FAPI-46 tracer uptake (SUV max, SUVmean and SUVpeak) in primary tumour, lymph node and distant metastases and background uptake in a dynamic scan protocol (expressed in Standardised Uptake Values).
Blood activity measurements of [68Ga]Ga-FAPI-46 tracer | 3 months
  [68Ga]Ga-FAPI-46 blood activity concentration (expressed in kBq/ml)
Plasma to blood ratio of [68Ga]Ga-FAPI-46 tracer | 3 months
  [68Ga]Ga-FAPI-46 plasma to blood ratio (expressed in kBq/ml)
Repeatability | 3 months
  The daily variability (average percentage of difference) of the preferred simplified method for quantification of [68Ga]Ga-FAPI-46.
Diagnostic accuracy | 3 months
  Per lesion analysis of diagnostic accuracy of [68Ga]Ga-FAPI-46 PET/CT using visual, semi quantitative and histopathological results.
Response monitoring | 3 months
  Accuracy of response monitoring of neoadjuvant therapy using [68Ga]Ga-FAPI-46 PET/CT in comparison to conventional imaging and histopathological results.

SECONDARY OUTCOMES:
Agreement imaging and pathology | 3 months
  Percentage of agreement between tumor uptake on the [68Ga]Ga-FAPI-46 PET/CT scan, histopathologic evidence of tumor, and the expression of FAP (IHC).
Agreement imaging modalities | 3 months
  Percentage of agreement between different imaging modalities ([68Ga]Ga-FAPI-46 PET/CT and CT , MRI or FDG PET/CT).
Imaging and tumor regression | 3 months
  Correlation between [68Ga]Ga-FAPI-46 PET/CT signal to tumor regression (MDACC method).
Change of therapy management | 3 months
  Percentage of potential change of therapy management enabled by [68Ga]Ga-FAPI-46 PET/CT.
Response prediction first scan | 3 months
  Sensitivity of response prediction of neoadjuvant therapy based on the first [68Ga]Ga-FAPI-46 PET/CT.
Resectability (based on DPCG criteria) | 3 months
  Accuracy of determining surgical resectability, based on DPCG criteria, using [68Ga]Ga-FAPI-46 PET/CT.
Diagnostic accuracy of incidental findings | 3 months
  Determine the diagnostic accuracy of incidental findings on [68Ga]Ga-FAPI-46 PET/CT using other imaging modalities, histopathological results, biopsy results, follow-up or a combination of the previous.

CONTACTS AND LOCATIONS:
Overall Officials: Rutger-Jan Swijnenburg, MD, PhD, Principal Investigator — Amsterdam UMC, location AMC
Locations (1):
- Amsterdam UMC, location VUmc, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be shared anonymously only of the participants who have given informed consent to share their data for other research proposes.
Supporting Information: Study Protocol, SAP
Time Frame: At the time of journal article publication.
Access Criteria: Research data may be provided upon a reasonable request with necessary privacy provisions and only data form participants who have given informed consent for the use data for other research.